CLINICAL TRIAL: NCT06834594
Title: Bleeding Patterns in Sequential and Continuous Progesterone Supplementation in Adolescents With Turner Syndrome: A Non-randomized Prospective Trial (The BOOST Study)
Brief Title: Bleeding Patterns in Sequential and Continuous Progesterone Supplementation in Adolescents With Turner Syndrome
Acronym: BOOST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003252
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Turner Syndrome; Primary Ovarian Insufficiency (Poi)
Keywords: Turner syndrome; Primary ovarian insufficiency; Hormone replacement therapy
MeSH Terms: conditions — Turner Syndrome; Primary Ovarian Insufficiency | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequential progesterone supplementation (Active Comparator): Oral micronized progesterone 200mg for the first 12 days of a 30 to 31-day cycle.
  Interventions: Drug: Micronized progesterone 200 MG
- Continuous progesterone supplementation: (Active Comparator): Oral micronized progesterone 100mg daily taken throughout the 30 to 31-day cycle.
  Interventions: Drug: Micronized Progesterone 100 MG

INTERVENTIONS:
Drug: Micronized progesterone 200 MG — Oral micronized progesterone 200mg for the first 12 days of a 30 to 31-day cycle
  Other Names: Sequential
  Arms: Sequential progesterone supplementation
Drug: Micronized Progesterone 100 MG — Oral micronized progesterone 100mg daily taken throughout the 30 to 31-day cycle.
  Other Names: Continuous
  Arms: Continuous progesterone supplementation:

SUMMARY:
This is a single-site open label non-randomized study comparing effects of sequential versus continuous use of progesterone supplementation amongst Turner Syndrome (TS) patients with primary ovarian insufficiency (POI) prescribed hormone replacement therapy (HRT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Turner Syndrome and Primary Ovarian Insufficiency.
* Prescribed adult dosing* of transdermal or oral estradiol for estrogen replacement therapy.

  *Adult dosing of will be defined per published clinical practice guidelines from the 2023 International Turner Syndrome Meeting (i.e. 50-200μg/day of transdermal estradiol, or (i.e. 50-200μg/day of transdermal estradiol or 2-4mg/day oral estradiol).
* Have achieved menarche.

Exclusion Criteria:

* Disclosure of sexual activity and desire for contraception.
* Having a levonorgestrel-releasing intrauterine device or etonogestrel arm implant in place.
* Having received depot medroxyprogesterone within one year prior to study recruitment.
* Non-English or non-Spanish speaking.

Ages: 12 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Menstrual bleeding patterns as assessed by the Pictorial Bleeding Assessment Chart (PBAC) | From enrollment to end of treatment at day 90.
  PBAC is one of the most common scoring systems used in the literature to quantify menstrual blood loss (MBL) using a pictorial scoring system, with a higher score representing a larger MBL and a score >100 qualifying as heavy menstrual bleeding

SECONDARY OUTCOMES:
Menstrual distress questionnaire (MEDI-Q) | From enrollment to end of treatment at day 90.
  The Menstrual distress questionnaire (MEDI-Q) is a valid and reliable instrument for the assessment of menstrual distress and its impact on psychological well-being. This tool can be utilized in research and clinical settings to comprehensively investigate the impact of menstruation on various populations
Endometrial thickness. | On study day 90 +/- 14 days.
  Endometrial thickness measured by transabdominal pelvic ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Tazim Dowlut-McElroy, M.D., M.S., Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Protect confidentiality of individuals with this rare disease (Turner syndrome).

REFERENCES:
- [Background] Gravholt CH, Andersen NH, Christin-Maitre S, Davis SM, Duijnhouwer A, Gawlik A, Maciel-Guerra AT, Gutmark-Little I, Fleischer K, Hong D, Klein KO, Prakash SK, Shankar RK, Sandberg DE, Sas TCJ, Skakkebaek A, Stochholm K, van der Velden JA; International Turner Syndrome Consensus Group; Backeljauw PF. Clinical practice guidelines for the care of girls and women with Turner syndrome. Eur J Endocrinol. 2024 Jun 5;190(6):G53-G151. doi: 10.1093/ejendo/lvae050. PMID 38748847
- [Background] Panay N, Anderson RA, Bennie A, Cedars M, Davies M, Ee C, Gravholt CH, Kalantaridou S, Kallen A, Kim KQ, Misrahi M, Mousa A, Nappi RE, Rocca WA, Ruan X, Teede H, Vermeulen N, Vogt E, Vincent AJ; ESHRE, ASRM, CREWHIRL, and IMS Guideline Group on POI. Evidence-based guideline: premature ovarian insufficiency. Hum Reprod Open. 2024 Dec 9;2024(4):hoae065. doi: 10.1093/hropen/hoae065. eCollection 2024. PMID 39660328
- [Background] Dowlut-McElroy T, Kanakatti Shankar R. Hormone Replacement Therapy after Pubertal Induction in Adolescents and Young Adults with Turner Syndrome: A Survey Study. Horm Res Paediatr. 2024;97(1):62-69. doi: 10.1159/000530724. Epub 2023 Apr 24. PMID 37094554
- [Background] Dowlut-McElroy T, Shankar RK. The Care of Adolescents and Young Adults with Turner Syndrome: A Pediatric and Adolescent Gynecology Perspective. J Pediatr Adolesc Gynecol. 2022 Aug;35(4):429-434. doi: 10.1016/j.jpag.2022.02.002. Epub 2022 Mar 8. PMID 35272055